CLINICAL TRIAL: NCT05583214
Title: Comparing the Efficacy of Ondansetron, Dexamethasone, and Placebo for the Reduction of Intraoperative Nausea and Vomiting in Patients Undergoing Lower-segment Caesarean Section Under Spinal Anesthesia
Brief Title: Evaluating the Effectiveness of Ondansetron Versus Dexamethasone Versus Placebo for the Control of Intraoperative Nausea and Vomiting in Patients Undergoing Lower-segment Caesarean Section Under Spinal Anesthesia
Acronym: ODP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Muhammad Mubariz (Other)
Responsible Party: Sponsor-Investigator, Muhammad Mubariz, House Officer, Akhtar Saeed Medical and Dental College
Organization: Akhtar Saeed Medical and Dental College (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UMO708991
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Caesarean Section; Spinal Anesthesia
MeSH Terms: interventions — Ondansetron; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ondansetron (Experimental): Patients given Ondansetron (8mg)
  Interventions: Drug: Ondansetron 8mg
- Dexamethasone (Experimental): Patients given Dexamethasone (8mg)
  Interventions: Drug: Dexamethasone 8mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ondansetron 8mg — 8mg of Ondansetron IV stat will be given to the group after induction of spinal anesthesia
  Arms: Ondansetron
Drug: Dexamethasone 8mg — 8mg of Dexamethasone IV stat will be given to the group after induction of spinal anesthesia
  Arms: Dexamethasone
Drug: Normal saline — Normal saline will be given IV stat to the group after induction of spinal anesthesia
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of Ondansetron, Dexamethasone, and Placebo for intraoperative nausea and vomiting in patients undergoing caesarian section under spinal anesthesia. The main question it aims to answer are:

Which drug is the best at reducing the incidence of intraoperative nausea and vomiting.

Which drug is the best at reducing intraoperative pain.

Participants will be randomly divided into three groups, each will be given a different drug labelled A, B, or C.

A rating scale will be used to evaluate the severity of intraoperative nausea and pain. Episodes of vomiting will be recorded.

Data collected from the three groups will be analyzed using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Age above 20 but less than 35 years old
* Given informed consent
* No contraindication to spinal anesthesia
* ASA I or II

Exclusion Criteria:

* Age less than 20 or more than 35 years old
* Non-consenting
* Contraindication to spinal anesthesia
* ASA III or IV

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative nausea | 20 minutes after initiation of procedure
  Measured by an 11-point numeric rating scale
Intraoperative vomiting | 1 hour
  Number of episodes of vomiting throughout the procedure

SECONDARY OUTCOMES:
Intraoperative pain | 20 minutes after the initiation of procedure
  Measured by an 11-point numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Mubariz, MBBS, Principal Investigator — House Officer
Locations (1):
- Akhtar Saeed Trust Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Patient's consent form, MR number Detailed rating scale data Intraoperative blood pressure and heart rate data
Supporting Information: Study Protocol, SAP, CSR